CLINICAL TRIAL: NCT04635514
Title: Lateral Colporrhaphy - a New Surgical Intervention: Case Series Study
Brief Title: Lateral Vaginal Wall Site-specific Defect Reconstructions
Status: Completed | Type: Observational
Sponsor: Institute of Gynecology, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IGynecology
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Gynecological Disorder
Keywords: Lateral vaginal wall anatomy; Lateral colporrhaphy
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group of 32 subjects: Thirty-two women who presented with symptomatic lateral vaginal prolapse (deep dyspareunia, sensation of vaginal fulness, and heaviness) composed the study's group.
  The surgical lateral vaginal reconstruction (lateral colporrhaphy) of the lateral vaginal wall was administered.
  Interventions: Procedure: Lateral colporrhaphy

INTERVENTIONS:
Procedure: Lateral colporrhaphy

SUMMARY:
LATERAL COLPORRHAPHY: A NEW SURGICAL INTERVENTION:

CASE SERIES STUDY

Background The surgical anatomy of site-specific defects of lateral vaginal wall (LVW) prolapse into the canal and its treatment are described for the first time.

Materials and Methods Thirty-two women who presented with symptomatic LVW prolapse (deep dyspareunia, sensation of vaginal fulness, and heaviness) were study. Before surgery, gross anatomy and the lateral colporrhaphy rehearsals had been performed on ten-human fresh female cadavers. A case series study was designed and conducted. Objectives were to ascertain the surgical anatomy within lateral vaginal wall site-specific defects; to evaluate whether lateral colporrhaphy can cure or improve symptoms; to describe a new lateral colporrhaphy. The primary outcome measured occurrences of site-specific defects within the lateral vaginal wall. The secondary outcome measured objective and subjective cure rates of lateral colporrhaphy.

Results Twenty-eight women (87.5%) concluded the study. The mean age of women was 46 ± 12 years, BMI 26.7 ± 2 kg/m2, and vaginal parity 2 ± 1. In all subjects, LVW defects had bulged into the vaginal canal. Lateral colporrhaphy yielded objective and subjective cure rates of 93% and 97%, respectively. Symptomatic improvements were recorded in 7%. The LVW surgical anatomy consisted of the full thickness of the vaginal wall, pubovaginalis muscle with fascia, and the perineal membrane.

Conclusions Symptomatic site-specific defects occur within the lateral vaginal wall. Lateral colporrhaphy cures or improves symptoms in this study group. The new lateral colporrhaphy procedure is a simple surgical intervention and is easy to perform.

DETAILED DESCRIPTION:
Material & methods

2.1 Ethics The author follows the ethical standards in this clinical-scientific study and complains with the Declaration of Helsinki [7, 8]. The local Institutional Review Board (IRB) was consulted with the study protocol and informed consent. Based on the Declaration of Helsinki, Section C, entitled "Unproven Interventions in Clinical Practice," the study was excluded from an IRB formal process. IRB advised referencing the Helsinki Declaration [7, 8]. All subjects had been furnished with informed consent in writing before enrollment. The cadaver study was approved by the local university Ethics Committee (no. AKBE 146/12).

2.2 Preoperative Evaluation The Numeric Pain Rating Scale (NPRS) was used to determine the severity of dyspareunia, and the subject's report was incorporated in evaluating other symptoms. All study participants were furnished with the standardized self-reported (NPRS) form. The numeric formula ranging from 0 to 10 (0, no pain; 1- 4, mild pain; 5 -7, moderate pain; 8-10, severe pain). Patients' dyspareunia severity was recorded based on the woman's real pain experience during vaginal intercourse.

The lateral vaginal walls were assessed from fornix to the exterior vaginal introitus, site-specific defects were identified and recorded, and photos were taken. Deep dyspareunia was reproduced during a clinical vaginal evaluation by poking a defective lateral vaginal wall. Induced surrogate pain was the endpoint for actual in-depth deep dyspareunia evaluation. In each follow-up visit, the author determined the objective cure rate with patient assistance. For this purpose, Extra-Absorbent Large Tipped Applicators with Plastic Handle (Puritan Medical Products, Guilford, ME 04443-0149, USA) were used. Patients reported the severity of pain, and the author charted pain. The protruding part of the LVW into the vaginal canal was evaluated by direct visualization. The prolapsing part was measured from the base of LVW to the most protruded portion of the lateral vaginal. This evaluation was applied preoperatively and during each follow-up visit.

2.3 Data Collection and Analysis Objective data were collected during a one-on-one interview performed by the author with every subject. Subjective data collected before and after surgery and yearly intervals until the completion of the follow-ups. Findings were compared with preoperative results, follow-up visits, and recorded.

2.4 Literature Search Zotero - reference manager, and PubMed, and other non-indexed studies were used for electronic medical literature searches regarding the lateral vaginal wall anatomy, site-specific defects within this structure, and surgical reconstruction. The Medical Subject Headings (MeSH) applied to gather relevant articles. Conference Proceedings and specializing website included in searches. Keywords were used: Vaginal wall anatomy; Vaginal wall surgical anatomy; Vaginal wall defects; Vaginal introitus; Vaginal tightening; Vaginal introitus; Vaginal walls; Lateral vaginal wall defects; Lateral vaginal wall defect repairs; Vaginal colporrhaphy.

2.5 Informed Consent Every subject in the before enrollment received written informed consent, which is presented in the present study. At the time of pre-surgical consultation, all patients were educated, in understandable terms, on the lateral colporrhaphy. The formal inform consent is included in the supplemental file.

2.6 Local Anesthesia All lateral colporrhaphy performed under local anesthesia. One-hour before the operation, a mixture of Lidocaine/Prilocaine (2.5%/2.5%) cream would be applied by the patient to the vaginal canal, the posterior perineum, the vaginal vestibule. Thirty minutes before the surgery, orally, Valium 2.5-5 mg and Phenergan 12.5 mg rectal suppository for light conscious sedation was administered. Bupivacaine 0.5 % with epinephrine solution (Hospira, Inc., Lake Forest, IL USA) used for vaginal wall infiltration if a patient was not sensitive to this agent (a skin test would be done before a surgical intervention).

2.7 Inclusion and Exclusion Criteria The consecutive corpses who demised within 24-hour and did not undergo a preservation process were included for the study and rehearsal. Those alive women who presented with lateral vaginal defects prolapsing into the vaginal canal and affiliated with moderate to severe deep dyspareunia were included. Anteverted uterus, anterior or posterior, colporrhaphy, and intact paravaginal suspension were prerequisites for inclusion. No concomitant procedure was performed during lateral vaginal wall repair. Women who presented with anterior or posterior vaginal wall defects (cystocele or rectocele), paravaginal defect, lateral vaginal defect, and did not have a prior surgical treatment for those conditions were excluded. Retroverted uterus, pregnancy, current infection of the lower genital tract, general illnesses, and inflammatory disorder constituted reasons for subjects being excluded from the study. Additionally, women who underwent a prior hysterectomy, bilateral oophorectomy, or had the diagnosis of vaginal dryness, endometriosis, prolapse, myofascial pain were excluded. A total of eight patients were excluded from the study.

2.8 Cadaveric Rehearsal Stratum-by-stratum anatomical cadaveric dissection was performed to verify the gross anatomy on one side of the same subject to identify the lateral vaginal wall and its supportive/suspending structures. On the other side of the same corps, rehearsal of the newly developed lateral vaginal wall colporrhaphy concept was exercised according to the narrative description of this surgical intervention, which is described below.

2.9 Surgical Intervention The surgery on live subjects was performed under x 3,5-4.0 magnifying loupe. A small vertical incision was made approximately 0.5 - 1.0 cm from the inner hymeneal ring on the lateral vaginal mucosa (between 2 and 3 o'clock on the left and 8 and 9 o'clock on the right side). The incision continued until after the full thickness of the vaginal wall was exposed. A traction suture, without tying, placed on the distal edge of the incision. The full thickness of the vaginal wall was dissected-off from vaginal inner-lateral defect. Approximately 1.0 cm above the proximal defect, another traction suture placed, without tying, and lateral sub-vaginal anatomical defect(s) was exposed. Both traction sutures were stretched, and scarification of defect edges was carried out until fresh oozing blood was observed. Edges of defects were approximated with a simple interrupted 2-0 delayed absorbable suture on a tapered, small needle. Site-specific defects reconstructions were completed in layers; the vaginal mucosa was trimmed and closed with a single interrupted 3-0 delayed stitch on a taper needle. Meticulous hemostasis was achieved. The overall procedure duration was measured in each case from the first incision to the operation's completion. The follow-up study was conducted at a one-year interval for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Those alive women who presented with lateral vaginal defects prolapsing into the vaginal canal and affiliated with moderate to severe deep dyspareunia were included. Anteverted uterus, anterior or posterior, colporrhaphy, and intact paravaginal suspension were prerequisites for inclusion.

Exclusion Criteria:

* Women who presented with anterior or posterior vaginal wall defects (cystocele or rectocele), paravaginal defect, lateral vaginal defect, and did not have a prior surgical treatment for those conditions were excluded. Retroverted uterus, pregnancy, current infection of the lower genital tract, general illnesses, and inflammatory disorder constituted reasons for subjects being excluded from the study. Additionally, women who underwent a prior hysterectomy, bilateral oophorectomy, or had the diagnosis of vaginal dryness, endometriosis, prolapse, myofascial pain were excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Thirty-two women who presented with symptomatic LVW prolapse (deep dyspareunia, sensation of vaginal fulness, and heaviness) composed the study. Before surgery, gross anatomy and the lateral colporrhaphy rehearsals had been performed on ten-human fresh female cadavers. A case series study was designed and conducted.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-11-15 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Occurrences of site-specific defects within the lateral vaginal wall | Duration of the surgical phase of the study
  To determine the existing of defects during actual surgery

SECONDARY OUTCOMES:
Measuring objective and subjective cure rates of lateral colporrhaphy. | Duration of the surgical phase of the study
  A lateral colporrhaphy performed per the study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ostrzenska, Study Director — Institute of Gynecology, Inc.

IPD SHARING:
Plan to Share IPD: Undecided